CLINICAL TRIAL: NCT07018726
Title: Addressing Emotional Distress in Dyads of Persons With a Young Onset Dementia (YOD) and Their Care-partners
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Full Professor/Director, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025P001534
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Young Onset Dementia
Keywords: Emotional Distress; Dyadic Intervention; Young Onset Dementia; Caregiving

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Experimental Patient-Caregiver Dyads (Experimental): There will be 6 sessions delivered via live video using Zoom. Content will be primarily skills.
  Interventions: Behavioral: Resilient Together-YOD
- Control Patient-Caregiver Dyads (Active Comparator): There will be 6 sessions delivered via live video using Zoom. Content will be primarily educational.
  Interventions: Behavioral: Health Enhancement Program-YOD

INTERVENTIONS:
Behavioral: Resilient Together-YOD — This is a 6 session dyadic (patient and spousal care-partner) intervention that teaches resiliency and interpersonal communication skills early after YOD diagnoses. It aims to decrease heightened symptoms of depression and anxiety among dyads to help them engage in important decisions around long term care-planning and optimize adjustment. The goal is to equip dyads with the necessary skills to cope and engage in meaningful, challenging conversations around care-planning, symptom deterioration, work/family planning to improve well-being in both members of the dyad.
  Other Names: Skills-based intervention
  Arms: Experimental: Experimental Patient-Caregiver Dyads
Behavioral: Health Enhancement Program-YOD — This is a 6 session program that will deliver educational information to dyads and will mimic the dose and duration of Resilient Together. The program will not teach any individual and dyadic interpersonal skills, but will contain education on psychological distress and healthy behaviors. Sessions will also be delivered virtually.
  Other Names: Educational program
  Arms: Control Patient-Caregiver Dyads

SUMMARY:
The purpose of the present investigation is to test the efficacy of a virtual, brief (6 sessions) dyadic (patient and care-partner together) intervention to prevent chronic emotional distress in dyads where one person is diagnosed with Young Onset Dementia (YOD). Through this study, we seek to address the unmet need of preventing chronic emotional distress in YOD dyads through a feasible, acceptable and credible program, and ideally enhance resiliency and improve wellbeing and quality of life in both members of the dyad.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 at the time of enrollment [both patient and care-partner]
* Diagnosis of young-onset dementia (FTD, PPA, AD, PCA, etc.) with symptom onset prior to age 65 [patient]
* A designated care-partner willing and interested to participate [both patient and care-partner]
* Received YOD diagnosis in the past 6 month [patient]
* English fluency and literacy [both patient and care-partner]
* Cognitive ability to understand study and research protocol in order to consent to study participation per referring neurologist [both patient and care-partner]
* Patient and/or caregiver exhibit emotional distress on screening (using HADS D and/or HADS A scores > 7)

Exclusion Criteria:

* An additional, terminal diagnosis such as cancer
* Lack of access to internet and/or a device with a camera
* Current untreated or unstable severe mental health conditions like bipolar disorder, schizophrenia, or active substance use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Emotional Distress | 0 weeks, 6 weeks, 12 weeks
  Hospital Depression and Anxiety Scale total score (HADS); 0-21 for each subscale (anxiety and depression), higher scores indicate greater anxiety or depression

SECONDARY OUTCOMES:
Change in Resiliency Factors (Mindfulness) | 0 weeks, 6 weeks, 12 weeks
  Cognitive and Affective Mindfulness Scale (CAMS); 12-48, higher scores indicate greater perceived mindfulness
Change in Resiliency Factors (Individual Coping) | 0 week, 6 weeks, 12 weeks
  Measure of Current Status Part A (MOCS-A) Assertiveness and Coping Confidence subscales; Subscale scores: 0-4; higher scores indicate greater perceived ability to cope
Change in Resiliency Factors (Mindfulness Utilization) | 0 weeks, 6 weeks, 12 weeks
  Applied Mindfulness Scale (AMPS); 0-60, higher scores indicate greater use of mindfulness practices.
Changes in Interpersonal Factors (Dyad Coping) | 0 weeks, 6 weeks, 12 weeks
  Dyadic Coping Inventory (DCI); 37-185, higher scores indicate greater perceived coping in the context of a relationship
Changes in Resiliency Factors (Perceived Social Support) | 0 weeks, 6 weeks, 12 weeks
  Multidimensional Scale of Perceived Social Support (MSPSS); 12-84, higher scores indicate greater perceived social support from family, friends, and significant others
Changes in Resiliency Factors (Values-based Living) | 0 weeks, 6 weeks, 12 weeks
  Valuing Questionnaire (VQ); Progress and Obstruction Subscale Scores: 0-30, higher scores indicate living in greater accordance with one's values

OTHER OUTCOMES:
Global Impressions of Change | 6 weeks, 12 weeks
  Modified Global Impressions of Chance (MGIC); 1-7: Higher scores indicate greater perceived change in outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital (MGH), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No